CLINICAL TRIAL: NCT00948103
Title: Nitrous Oxide (KALINOX®) Inhalation and Tolerance of Intravesical Botulinum Neurotoxin A Injection: a Double-blind Randomized Controlled Study
Brief Title: The Interest of the Nitrous Oxide During Intravesical Injection of Botulinum Toxin A
Acronym: PROTOTOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P050701
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Injection Site Vesicles
Keywords: Nitrous Oxide; Administration, Intravesical Drug; Botulinum toxin
MeSH Terms: interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxygen (Placebo Comparator)
  Interventions: Drug: Oxygen
- Nitrous Oxide (Active Comparator)
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — nitrous oxide inhalation during intravesical injection. Dose depends on gender and pain
  Arms: Nitrous Oxide
Drug: Oxygen — oxygen
  Arms: Oxygen

SUMMARY:
Second line treatment for detrusor hyperreflexia is the intravesical BTX-A injections. First 300 units Botox are diluted with 30 ml of preservative-free saline. Using a rigid cystoscope and an injection needle, BTX-A is injected into 30 sites within the detrusor muscle.

The used of KALINOX® (50% nitrous oxide and oxygen) inhalation has demonstrated analgesic efficacy in various procedures (obstetric, liver biopsy, transrectal ultrasound guided prostate biopsy, emergency) The aim of this study is to investigate the safety and efficacy of analgesia with N2O/O2 inhalation for detrusor BTX-A injections using a rigid cystoscope.

DETAILED DESCRIPTION:
First line treatment for detrusor hyperreflexia is the use of antimuscarinic medications. However, these medications can have unwanted side effects and often are not good enough to decrease incontinence in cases of severe neurogenic detrusor overactivity. Some invasive surgical procedures are possible such as sacral nerve stimulator, sacral rhizotomy, bladder myomectomy and bladder augmentation. But there are still few treatment option for this medical complication. Recently, some data are showed the clinical application of botulinum neurotoxin A (BTX-A) into detrusor muscle in cases of resistant neurogenic detrusor overactivity to conventional treatment with anticholinergic medication. In these studies the authors perform intravesical BTX-A injections. First 300 units Botox are diluted with 30 ml of preservative-free saline. Using a rigid cystoscope and an injection needle, BTX-A is injected into 30 sites within the detrusor muscle.

To reduce the pain, instillation of lidocaine before botulinum-A toxin injections is used into the bladder. On a 10-point rating scale the mean pain score of the patients who underwent the injections of Botox after conventional lidocaine instillation is 4.0 (SD 1.6).

The used of KALINOX® (50% nitrous oxide and oxygen) inhalation has demonstrated analgesic efficacy in various procedures (obstetric, liver biopsy, transrectal ultrasound guided prostate biopsy, emergency…) associated with mild to moderate pain and it is technically simple to use. Early studies indicated that 30% nitrous oxide is equipotent to 10 to 15 mg. morphine. Except in patients with severe chronic obstructive pulmonary disease KALINOX® inhalation is a safe and acceptable method of sedation and analgesia. It is a nonirritant and is excreted unchanged from the lungs.

The aim of this study is to investigate the safety and efficacy of analgesia with N2O/O2 inhalation for detrusor BTX-A injections using a rigid cystoscope. Will be included patient with severe neurogenic detrusor overactivity but with preserved bladder sensibility treated with botulinum-A toxin injections into the detrusor muscle Patients will be randomized into a group that will receive KALINOX® via a breath activated device and a control group that receive oxygen through a similar breathing device. The investigator will be involved in the randomization process since the gas cylinders will be covered and they will be blind to the gas used. All patients involved will be blinded to the gas that they will inhale. The patients will score the injection pain and the anxiety on a 10-point rating scale. Furthermore the duration of the practice will be measured.

The hypothesis is that analgesia with KALINOX® will show a significant difference in pain perception among the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman of more than 18 years
* Patient with overactive bladder
* First intravesical Botulinum injection
* Bladder sensitivity on the urodynamic
* Patient not presenting contraindication to this injection
* Cystoscopy realized before the injection of botulinal toxin A
* Negative pregnancy test for women of child-bearing age
* Signing of an informed consent form, after appropriate information has been provided

Exclusion Criteria:

* Pregnancy
* Contraindication in the toxin such as severe myasthenia, syndrome of Eaton-Lambert, or amyotrophic lateral sclerosis
* Treatment antibiotic by aminoglycoside
* Allergies known about the toxin, about the anesthetics used during the study
* Patients under anticoagulants, or having taken a treatment anti-aggregant platelet in 10 days preceding the injection
* Haemophilia or deficit in factor of the coagulation responsible for disorder of the haemostasis
* Current urinary infection defined in the ECBU by a superior bacteriuria in 10°5 / ml and a leucocyturia superior to 10°4 / ml
* Current genital infection or in four weeks preceding the injection
* Histories of irradiation pelvic or treatment in the course of a neoplasia
* Current treatment or in six months preceding the randomisation by a pharmacological ENDOVESICAL agent
* Patients requiring a ventilation in pure oxygen
* Intra-cranial high blood pressure
* Conscience alteration
* Lung diseases
* Bubbles of emphysema
* Gaseous embolism
* Accident of dive
* Abdominal gaseous distension
* Patient having received recently an ophthalmic gas (SF6, C3F8, C2F6) used in the eye surgery as long as persists a bubble of gas inside the eye and at least during a period of 3 months
* Facial traumatism
* Chronic respiratory failure
* Analgesic treatment by morphine or morphine agonists of class 3
* Psychiatric pathology interfering with the compliance to the protocol or not allowing a correct evaluation of the result
* Patient having participated in a clinical study in 3 months preceding the inclusion
* No affiliation to any social insurance system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mean pain during intravesical injection | 5 minutes

SECONDARY OUTCOMES:
Maximum pain during intravesical injection | 5 minutes
Anxiety during intravesical injection | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DENYS, PUPH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Raymond Poincaré, Garches, France